CLINICAL TRIAL: NCT02729662
Title: Longitudinal Efficacy and Safety Study of Tolvaptan on Autosomal Dominant Polycystic Kidney Disease Patients (LET-PKD Study)
Brief Title: Efficacy of Tolvaptan on ADPKD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Eiji Higashihara, MD, Adjunct Professor, Kyorin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LET-PKD-1
Record Dates: First submitted 2016-03-11; First posted 2016-04-06 (Estimated); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with ADPKD (Other): This analysis set consists of patients whose at least 2 TKV data are available both before and after taking tolvaptan.
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan — * Before administration of tolvaptan
    * TKV・Liver capacity: Once/year (an additional measurement within 3 months before start of administration)
    * 24-hour urine collection・Hematology/urinalysis: Once/year
    * Physical findings: Blood pressure and medical interview at ambulatory visit
  * Hospitalization for education and examination at the start of tolvaptan administration
    * 24-hour urine collection・Hematology/urinalysis・Inulin clearance
    * Physical findings: Body weight, blood pressure
    * Adverse Events
  * After administration of tolvaptan
    * TKV・Liver capacity・inulin clearance: Once/year
    * 24-hour urine collection: Once/6 months
    * Hematology/urinalysis: Once/month in principle
    * Physical findings: Blood pressure and medical interview at ambulatory visit
    * Adverse Events
  Other Names: Samsca

SUMMARY:
Investigation of the therapeutic effects of tolvaptan in patients with autosomal dominant polycystic kidney disease This is a prospective 5-year study to compare the change in total kidney volume (TKV) before and after tolvaptan therapy, as the primary endpoint, in patients with ADPKD. Study results will be summarized, analyzed, and compiled into a research paper at 5 years (data cut-off, Aug 31, 2020).

DETAILED DESCRIPTION:
Based on the results of a study entitled "The Tolvaptan Efficacy and Safety in Management of Autosomal Dominant Polycystic Kidney Disease and Its Outcomes (TEMPO 3:4) 1)," tolvaptan was approved in March 2014 for the treatment of autosomal dominant polycystic Kidney Disease (ADPKD) in Japan, followed by in other regions such as Europe and Canada.

In May 2014, Kyorin University Hospital started administration of tolvaptan to patients with ADPKD. In the clinical setting in which the dosing conditions differ from those in the TEMPO study, aspects that were not addressed in the TEMPO study may be investigated. The present study is a longitudinal clinical study to investigate the changes before and after administration of tolvaptan by employing a method different from that used in the TEMPO study in patients in whom the clinical course of the disease has been monitored since prior to the approval of tolvaptan.

The observation period (for a maximum duration of 3 years) of the study was originally planned to be completed on March 31, 2018 and the analyses of study results and the preparation of a research paper until September 2019. However, the study will be extended for another 2 years, because the long-term effects of the drug should be further investigated.

The indication approved in Japan defines the target population as those with an eGFR ≥15 mL/min/1.73 m2, but not specifies the upper limit of age. Therefore, the present study will permit the assessment of therapeutic effects of the drug in patients who are older or have more severe renal impairment as compared with in those participating in the TEMPO3:4 and 4.4 studies. Since such patients generally have a greater TKV, the study may also provide information to decide whether the efficacy of tolvaptan differs according to TKV. The present study is a single-arm longitudinal study, unlike the preceding studies that were placebo-controlled studies 1,2); therefore, tolvaptan may be evaluated from different perspectives.

Rationale of DNA analysis The association between pathogenic genotype and the effects of tolvaptan has been reported, but the impact of mutation site has not been cleared 2). Genetic analysis for polycystic kidney will be included in the study to decide whether the effects of tolvaptan is associated with mutation site as well as pathogenic genotype (PKD1, PKD2).

Validation of alpha as a HtTKV slope Assuming that TKV corrected for the height at the age at measurement (t years old), HtTKVt (mL/m), increases at a constant annual rate (α, %/ per year) and the HtTKV0 is 150 mL/m, the following equation will be satisfied: HtTKVt = 150 (1+α)t. The α value calculated from the equation will be used as an indicator for supplementarily assessing the effect of tolvaptan on HtTKV slope 5,6).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have started or will start receiving tolvaptan at Kyorin University Hospital.
2. Patients whose use of Samsca complies with the criteria specified by the Ministry of Health, Labour and Welfare.

   * TKV ≥ 750 mL.
   * The increase in total renal capacity ≥ approximately 5%/year.
3. Patients who have given signed consent to the examination protocol, which includes hospitalization at the initiation of tolvaptan treatment (i.e. examination/educational hospitalization for the first 3 days. Monthly blood tests at the time of ambulatory visits, 24-hour urine collection every 6 months, annual TKV measurement by MRI and inulin clearance measurement)
4. Patients for whom the baseline TKV and eGFR percent change is available.
5. Patients from whom freely given, written informed consent to participate in the study has been obtained.

Exclusion Criteria:

1. Patients who do not consent to participation in the study, or those who later withdraw their consent.
2. Patients who have been taking tolvaptan since the TEMPO study.
3. Patients who are not eligible at our hospital to take tolvaptan for the stated indication based on the criteria for careful administration of Samsca as specified by the Ministry of Health, Labour and Welfare.

   * Patients with a history of hypersensitivity to tolvaptan or similar chemical compounds.
   * Patients who do not feel thirsty or have difficulty swallowing water.
   * Patients with hypernatremia.
   * Patients with eGFR < 15 mL/min/1.73 m2.
   * Patients with chronic hepatitis, drug-induced hepatic dysfunction and other hepatic dysfunctions.
   * Pregnant women or women suspected of being pregnant. Female patients who wish to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
The percent change in TKV volumetrically | once a year, up to study completion, an expected average of up to 5 years
  To evaluate the efficacy, the percent change in TKV volumetrically measured by MRI (% per year) is to be compared before and after administering tolvaptan to the same patients. The evaluation will include stratified analyses by patient background variables and examination data obtained during treatment.
  [Supplementary assessment of the primary outcome variable] Using HtTKV slope, α (% per year), calculated from the HtTKVt at t years old as an indicator, the effect of tolvaptan on HtTKV slope will be supplementarily assessed 5,6).

SECONDARY OUTCOMES:
The percent change in epidermal growth factor receptor (eGER) | once a month, up to study completion, an expected average of up to 5 years
  The percent change in eGFR (mL/min/1.73 m2 per year) will be compared before and after administration for evaluation. The evaluation will include stratified analyses by patient background variables and examination data obtained during treatment.
A number of adverse events during the study | through study completion, an expected average of up to 5 years
  The following events that occurred in subjects who received a medicinal product of Otsuka Pharmaceutical from the time of informed consent and in the time of the study completion will be recorded.
  1. Serious adverse event
  2. Non-serious adverse event
  3. Pregnancy
  4. Other safety information
The efficacy of or response to tolvaptan will be evaluated. | twice a year, up to study completion, an expected average of up to5 years
  Based on the data obtained from 24-hour urine collection (Urine volume, urinary protein, Na, K, Cl, UN, creatinine, NAG, β2-MG, albumin, urinary osmolality), blood tests (Na, K, Cl, Ca, IP, BUN, creatinine, eGFR, uric acid, total protein, albumin, globulin, total bilirubin, γ-GTP, AST, ALT, HDL-cholesterol, LDL-cholesterol, triglyceride, cystatin-C, serum osmolality, WBC, RBC, Hb, Ht, Plt, MCV, MCH, MCHC, Retic), inulin clearance, and TKV, the efficacy of or response to tolvaptan will be evaluated. The evaluation will include stratified analyses by patient background variables, and examination data obtained during treatment.
The impact of tolvaptan on the correlation between inulin clearance and eGFR values | once a month, up to study completion, an expected average of up to 5 months
  The correlation between inulin clearance and eGFR values obtained from the formulae to estimate eGFR will be investigated to elucidate the impact of tolvaptan on the correlation.
The association between the result of DNA analysis and the effect of tolvaptan | through study completion, an expected average of up to 5 years
  The association between the result of DNA analysis and the effect of tolvaptan will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Eiji Higashihara, MD, Principal Investigator — Kyorin University School of Medicine
Locations (1):
- Kyorin University Hospital, Mitaka, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torres VE, Chapman AB, Devuyst O, Gansevoort RT, Grantham JJ, Higashihara E, Perrone RD, Krasa HB, Ouyang J, Czerwiec FS; TEMPO 3:4 Trial Investigators. Tolvaptan in patients with autosomal dominant polycystic kidney disease. N Engl J Med. 2012 Dec 20;367(25):2407-18. doi: 10.1056/NEJMoa1205511. Epub 2012 Nov 3. PMID 23121377
- [Background] Torres VE, Chapman AB, Devuyst O, Gansevoort RT, Perrone RD, Dandurand A, Ouyang J, Czerwiec FS, Blais JD; TEMPO 4:4 Trial Investigators. Multicenter, open-label, extension trial to evaluate the long-term efficacy and safety of early versus delayed treatment with tolvaptan in autosomal dominant polycystic kidney disease: the TEMPO 4:4 Trial. Nephrol Dial Transplant. 2017 Jul 1;32(7):1262. doi: 10.1093/ndt/gfx079. No abstract available. PMID 28444221
- [Background] Higashihara E, Nutahara K, Okegawa T, Shishido T, Tanbo M, Kobayasi K, Nitadori T. Kidney volume and function in autosomal dominant polycystic kidney disease. Clin Exp Nephrol. 2014 Feb;18(1):157-65. doi: 10.1007/s10157-013-0834-4. Epub 2013 Jul 18. PMID 23864346
- [Background] Higashihara E, Nutahara K, Okegawa T, Tanbo M, Hara H, Miyazaki I, Kobayasi K, Nitatori T. Kidney volume estimations with ellipsoid equations by magnetic resonance imaging in autosomal dominant polycystic kidney disease. Nephron. 2015;129(4):253-62. doi: 10.1159/000381476. Epub 2015 Apr 16. PMID 25895545
- [Background] Irazabal MV, Rangel LJ, Bergstralh EJ, Osborn SL, Harmon AJ, Sundsbak JL, Bae KT, Chapman AB, Grantham JJ, Mrug M, Hogan MC, El-Zoghby ZM, Harris PC, Erickson BJ, King BF, Torres VE; CRISP Investigators. Imaging classification of autosomal dominant polycystic kidney disease: a simple model for selecting patients for clinical trials. J Am Soc Nephrol. 2015 Jan;26(1):160-72. doi: 10.1681/ASN.2013101138. Epub 2014 Jun 5. PMID 24904092
- [Background] Girardat-Rotar L, Braun J, Puhan MA, Abraham AG, Serra AL. Temporal and geographical external validation study and extension of the Mayo Clinic prediction model to predict eGFR in the younger population of Swiss ADPKD patients. BMC Nephrol. 2017 Jul 17;18(1):241. doi: 10.1186/s12882-017-0654-y. PMID 28716055
- [Background] Kinoshita M, Higashihara E, Kawano H, Higashiyama R, Koga D, Fukui T, Gondo N, Oka T, Kawahara K, Rigo K, Hague T, Katsuragi K, Sudo K, Takeshi M, Horie S, Nutahara K. Technical Evaluation: Identification of Pathogenic Mutations in PKD1 and PKD2 in Patients with Autosomal Dominant Polycystic Kidney Disease by Next-Generation Sequencing and Use of a Comprehensive New Classification System. PLoS One. 2016 Nov 11;11(11):e0166288. doi: 10.1371/journal.pone.0166288. eCollection 2016. PMID 27835667
- [Background] Higashihara E, Horie S, Kinoshita M, Harris PC, Okegawa T, Tanbo M, Hara H, Yamaguchi T, Shigemori K, Kawano H, Miyazaki I, Kaname S, Nutahara K. A potentially crucial role of the PKD1 C-terminal tail in renal prognosis. Clin Exp Nephrol. 2018 Apr;22(2):395-404. doi: 10.1007/s10157-017-1477-7. Epub 2017 Oct 5. PMID 28983800
- [Background] Tan AY, Michaeel A, Liu G, Elemento O, Blumenfeld J, Donahue S, Parker T, Levine D, Rennert H. Molecular diagnosis of autosomal dominant polycystic kidney disease using next-generation sequencing. J Mol Diagn. 2014 Mar;16(2):216-28. doi: 10.1016/j.jmoldx.2013.10.005. Epub 2013 Dec 27. PMID 24374109
- [Background] Irazabal MV, Torres VE, Hogan MC, Glockner J, King BF, Ofstie TG, Krasa HB, Ouyang J, Czerwiec FS. Short-term effects of tolvaptan on renal function and volume in patients with autosomal dominant polycystic kidney disease. Kidney Int. 2011 Aug;80(3):295-301. doi: 10.1038/ki.2011.119. Epub 2011 May 4. PMID 21544064
- [Background] Boertien WE, Meijer E, de Jong PE, Bakker SJ, Czerwiec FS, Struck J, Oberdhan D, Shoaf SE, Krasa HB, Gansevoort RT. Short-term renal hemodynamic effects of tolvaptan in subjects with autosomal dominant polycystic kidney disease at various stages of chronic kidney disease. Kidney Int. 2013 Dec;84(6):1278-86. doi: 10.1038/ki.2013.285. Epub 2013 Jul 31. PMID 23903369